CLINICAL TRIAL: NCT00164372
Title: Collaborative Injection Drug Users Study III/Drug Users Intervention Trial (CIDUS III/DUIT)
Brief Title: Behavioral Intervention for HIV and HCV-Uninfected Injection Drug Users
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-2934; U64/CCU317662,; U64/CCU517656,; U64/CCU917655,; U64 CCU217659,; U64/CCU071615
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: HIV Infections; Hepatitis C
Keywords: IV Drug users; HIV; hepatitis C virus; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Peer Education Intervention

SUMMARY:
The purpose of this study is to test whether a six-session behavioral intervention for HIV and HCV seronegative injection drug users is effective in reducing sexual and injection risk behaviors that could lead to primary HIV and HCV infection.

DETAILED DESCRIPTION:
CIDUS III/DUIT is a five-city (Baltimore, Chicago, Los Angeles, New York, and Seattle) randomized controlled trial to develop and evaluate the efficacy of a six-session behavioral intervention for HIV and HCV uninfected injection drug users between the ages of 15 and 30 years. The primary goals of the intervention are to:

1. decrease the shared use of syringes and other injection paraphernalia,
2. decrease sexual risk behaviors associated with HIV and HCV infection, and
3. decrease the incidence of hepatitis C virus (HCV) infection.

The intervention arm consists of six small-group training and skills-building sessions to teach and reinforce peer education activities around decreasing sex and injection risk behaviors for HIV and HCV infection. In the fifth session, participants practice peer education around sex or injection risk behaviors within their community. The control arm consists of six video and discussion sessions to control for attention. Prior to study enrollment, all participants in both arms receive HIV and HCV testing with client-centered pre- and post-test counseling to also control for the demand for risk reduction information. Behavioral assessments (by audio computer assisted self interviewing) and blood draws (for serologic testing) occur at baseline, 3 and 6 month follow-up. 3285 participants completed the baseline visit, of whom 1564 tested HIV and HCV seronegative and returned for test results making them eligible to enroll in the intervention trial. Of the eligible participants, 854 were randomized into the trial. 606 and 591 returned for 3 and 6 month follow-up assessments, respectively, and 712 participants completed at least one follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* age 15-30 years old
* self-reported illicit drug injection within the past 6 months
* live in the geographic region under study and plan to stay for >12 months
* willing to provide a blood sample for serologic testing
* willing to provide basic contact information for follow-up
* able to communicate in English
* had not participated in the pilot study or previously enrolled in the trial
* not concurrently participating in other HIV or HCV intervention trials
* tested HIV and HCV seronegative at baseline

Exclusion Criteria:

-

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1400
Dates: Start 2002-05; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
1. decrease in the number and proportion of times participants practiced vaginal or anal sex without a condom.
2. decrease in the overall number of persons participants shared syringes or injection equipment with.
3. decrease in the number and proportion of injections done with a syringe previously used by another person.
4. decrease in the number and proportion of times participant used another person's equipment to prepare or divide drugs before injecting.

SECONDARY OUTCOMES:
1. decrease the incidence of HCV infection.
2. decrease the frequency of injecting in high-risk settings.
3. increase the frequency of drug treatment entry or decrease the frequency of injection drug use.

CONTACTS AND LOCATIONS:
Overall Officials: Richard S. Garfein, PhD, MPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (5):
- United States (5):
  - Health Research Association, Los Angeles, California
  - University of Illinois at Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - New York Academy of Medicine, New York, New York
  - Public Health Seattle and King County, Seattle, Washington

REFERENCES:
- [Derived] Mackesy-Amiti ME, Ouellet LJ, Golub ET, Hudson S, Hagan H, Garfein RS. Predictors and correlates of reduced frequency or cessation of injection drug use during a randomized HIV prevention intervention trial. Addiction. 2011 Mar;106(3):601-8. doi: 10.1111/j.1360-0443.2010.03251.x. Epub 2010 Dec 23. PMID 21182555
- [Derived] Garfein RS, Golub ET, Greenberg AE, Hagan H, Hanson DL, Hudson SM, Kapadia F, Latka MH, Ouellet LJ, Purcell DW, Strathdee SA, Thiede H; DUIT Study Team. A peer-education intervention to reduce injection risk behaviors for HIV and hepatitis C virus infection in young injection drug users. AIDS. 2007 Sep 12;21(14):1923-32. doi: 10.1097/QAD.0b013e32823f9066. PMID 17721100
- [Derived] Garfein RS, Swartzendruber A, Ouellet LJ, Kapadia F, Hudson SM, Thiede H, Strathdee SA, Williams IT, Bailey SL, Hagan H, Golub ET, Kerndt P, Hanson DL, Latka MH; DUIT Study Team. Methods to recruit and retain a cohort of young-adult injection drug users for the Third Collaborative Injection Drug Users Study/Drug Users Intervention Trial (CIDUS III/DUIT). Drug Alcohol Depend. 2007 Nov;91 Suppl 1:S4-17. doi: 10.1016/j.drugalcdep.2007.05.007. Epub 2007 Jun 19. PMID 17582705